CLINICAL TRIAL: NCT00213772
Title: "Factors Associated With Porphyria Cutanea Tarda in Patients Infected With Hepatitis C Virus"
Brief Title: Risk Factors of Porphyria Cutanea Tarda (PCT)
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Other Study IDs: 2030
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Porphyria Cutanea Tarda
Keywords: Porphyria cutanea tarda; hepatitis C; hemochromatosis
MeSH Terms: conditions — Porphyria Cutanea Tarda; Hepatitis C; Hemochromatosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Comparison of patients with documented PCT and HCV infection, documented PCT without HCV, HCV infection without PCT and controls without HCV or PCT.

Single blood + urine sample uptake to investigate : mutations in HFE gene, uroporphyrinogen decarboxylase activity, HCV genotye, history of disease.

ELIGIBILITY:
Inclusion Criteria:

* Porphyria cutanea tarda /HCV negative Porphyria cutanea tarda/ HCV positive HCV positive HCV negative controls

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cribier, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg; O. Chosidow, MD, Principal Investigator — Hopital Pitié-Salpétrière / Paris; M. Bagot, MD, Principal Investigator — Hopital Henri Mondor / CHU Créteil; J.P Lacour, MD, Principal Investigator — Hopital de l'Archet / CHU Nice